CLINICAL TRIAL: NCT06436846
Title: Characterization of the Genomic Risk Underlying Retroperitoneal Liposarcoma
Brief Title: Genomic Risk in Retroperitoneal Sarcoma
Status: Recruiting | Type: Observational
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 21-8008
Record Dates: First submitted 2024-05-07; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Retroperitoneal Liposarcoma; Soft Tissue Sarcoma
MeSH Terms: conditions — Retroperitoneal liposarcoma; Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples of retroperitoneal fat (x4), subcutaneous fat (x1), primary tumor samples (x3) - all collected during surgery for tumor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: The entire study is a singular cohort of patients with retroperitoneal liposarcoma (index or recurrent) who undergo surgical resection of their tumor.
  Interventions: Other: Biospecimen sample collection during standard-of-care surgery

INTERVENTIONS:
Other: Biospecimen sample collection during standard-of-care surgery — Patients in this observational study are undergoing planned surgical resection of their retroperitoneal sarcoma as prescribed by their primary surgeon and treatment team. In addition to removal of the primary tumor, surgeons remove 4 samples of retroperitoneal fat and a sample of subcutaneous fat for further study at the time of the operation.

SUMMARY:
The protocol intends to explore the biology which may underlie recurrences of retroperitoneal liposarcoma. Surgery remains the only curative intent intervention for this disease. Often, tumors recur in locations within the retroperitoneum remote from the original primary tumor. This study hypothesizes that normal appearing retroperitoneal fat actually harbors underlying genetic changes which predispose to development of future liposarcoma. To accomplish this goal, retroperitoneal fat is sampled from quadrants within and remote from the primary tumor and is subsequently subjected to genetic analyses looking for such predisposing factors.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥18 years).
* Histologically confirmed retroperitoneal liposarcoma via preoperative biopsy, or cross-sectional imaging suspicious for liposarcoma with planned surgical resection
* Will be undergoing surgical resection for treatment of primary or recurrent disease
* Have provided informed consent to participate in this study

Exclusion Criteria:

• Prior surgical anatomy which makes sampling of remote areas of the retroperitoneum technically impossible or clinically undesirable for safety reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients (age 18 years or older) with retroperitoneal tumors suspicious for liposarcoma.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Presence of MDM2 amplification in "normal" retroperitoneal fat | Through study completion, an average of 3 years
  MDM2 amplification of primary tumors and fat samples will be tested by immunohistochemistry and/or fluorescence in situ hybridization.

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No